CLINICAL TRIAL: NCT03554239
Title: Impact of Genotyping P450 2C19 on Hospitalization Period When Voriconazole Treatment is Started
Brief Title: Impact of Genotyping P450 2C19 on Hospitalization Period
Acronym: PHARMACOGEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/15/7853
Record Dates: First submitted 2016-09-07; First posted 2018-06-13 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Infection
Keywords: Genotyping techniques; Fungal infection
MeSH Terms: conditions — Infections; Mycoses | interventions — Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voriconazole treatment (Other): Patients who start voriconazole treatment and receive benefits of genotyping
  Interventions: Genetic: genotyping

INTERVENTIONS:
Genetic: genotyping — Blood sample

SUMMARY:
Monocentric study with the objective to evaluate the impact of genotyping CYP2C19 on the hospitalization period. The genotyping will permit to adapt at best the Voriconazole posology.

DETAILED DESCRIPTION:
The main objective of this multi-center study is to evaluate the impact of dose adjustment of Voriconazole after CYP2C19 genotyping at the start of treatment, on the length of hospital stay.

Thus, a new strategy will be proposed as part of this project and will be compared to the reference strategy:

The New strategy: genotyping of CYP2C19 in any patient receiving treatment with Voriconazole in order to better adapt the treatment regimen as quickly as possible (increase of the dosage of Voriconazole in high-speed metabolisers or use of another antifungal, decreased dosage in poor metabolisers).

The Reference strategy: pharmacological therapeutic monitoring of Voriconazole allowing an adaptation of the Voriconazole dosage based on the residual concentration measured once steady state has been reached (5 elimination half-lives).

Multicenter, randomized study comparing two strategies of Voriconazole adaptation according to whether or not genotyping of CYP2C19 is performed as soon as Voriconazole is started.

Thus, the new strategy tested in this project and compared to the reference strategy (adaptation of Voriconazole dosage depending on the residual concentration), will be a genotyping of CYP2C19 in any patient receiving a treatment based on Voriconazole in order to better adapt the treatment regimen as quickly as possible (increase in the dosage of Voriconazole or use of another antifungal agent in ultra-rapid metabolisers, decrease in dosage in poor metabolisers).

ELIGIBILITY:
Inclusion Criteria:

* Patient with Voriconazole treatment
* Man or woman
* With social security number

Exclusion Criteria:

* Patient or parent of patient who refuse to accept inform consent form
* All patient under protection of adults

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The length of stay hospitalization | 6 months
  This duration will be expressed in number of days and will be compared between patients who have been genotyped since the introduction of Voriconazole compared to patients who have received therapeutic monitoring of Voriconazole (reference strategy).

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Gandia, PharmD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided